CLINICAL TRIAL: NCT02173288
Title: Role of Midodrine and Tolvaptan in Patients With Cirrhosis With Refractory or Recurrent Ascites
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr.Virendra Singh, Professor of Hepatology, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Mido-tolvaptan 1
Record Dates: First submitted 2014-06-18; First posted 2014-06-24 (Estimated); Last update posted 2017-09-19 (Actual); Status verified 2017-09

CONDITIONS: Cirrhosis; Refractory/Recurrent Ascites
MeSH Terms: conditions — Fibrosis; Ascites | interventions — Furosemide; Tolvaptan; Midodrine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Standard medical therapy (Active Comparator): Standard Medical therapy (n-15) with100 to 400mg spironolactone and/or 40 to 160mg furosemide.
  Interventions: Drug: Standard medical therapy
- Midodrine group (Active Comparator): Standard medical therapy (n-15) with Midodrine 7.5 mg thrice a day
  Interventions: Drug: Standard medical therapy; Drug: Midodrine
- Tolvaptan group (Active Comparator): Standard medical therapy (n-15) with Tolvaptan 15 mg twice a day
  Interventions: Drug: Standard medical therapy; Drug: Tolvaptan
- Tolvaptan plus midodrine arm (Experimental): Standard medical therapy (n-15) with Tolvaptan 15 mg twice a day and Midodrine 7.5 mg thrice a day
  Interventions: Drug: Standard medical therapy; Drug: Tolvaptan; Drug: Midodrine

INTERVENTIONS:
Drug: Standard medical therapy
  Other Names: Standard Medical therapy (n-15) with100 to 400mg spironolactone and/or 40 to 160mg furosemide.
Drug: Tolvaptan
  Other Names: Tolvaptan 15 mg twice a day
  Arms: Tolvaptan group; Tolvaptan plus midodrine arm
Drug: Midodrine
  Other Names: Midodrine 7.5 mg thrice a day
  Arms: Midodrine group; Tolvaptan plus midodrine arm

SUMMARY:
The development of ascites in the natural history of cirrhosis heralds a worsening of the prognosis to 50% survival at 2 years, and this deteriorates to 30-50% at 1 year when the ascites becomes refractory to medical therapy. Hemodynamic alterations and their relation to neurohumoral systems are essential in pathophysiology of ascites formation. The theory that best explain the ascites formation and sodium retention in cirrhotics is portal hypertension leading to splanchnic arterial vasodilatation leading to underfilling of arterial circulation which is sensed by the arterial and the cardiopulmonary receptors leading to sympathetic nervous system activation and activation of the anti-natriuretic factors (RAAS and arginine vasopressin), resulting in sodium and water retention. The therapeutic options available for patients with refractory ascites are serial therapeutic paracentesis, liver transplantation and transjugular intrahepatic portosystemic shunts.Vasopressin V2 receptor antagonists antagonize the antidiuretic effects of vasopressin at the V2 receptor located in the renal collecting duct, they increase free water clearance, and thus may be helpful in mobilizing excess water in conditions associated with water retention including cirrhosis. The use of V2 receptor antagonists in cirrhosis with ascites has been shown to be safe and efficacious. Midodrine, an alpha adreno receptor agonist by causing splanchnic vasoconstriction has been used in hepatorenal syndrome (HRS) and for control of ascites in patients with refractory or recurrent ascites. It is possible that vasoconstrictors and aquaretics (V2 receptor antagonists) by acting at different sites in combination may reverse some of the pathogenic events that results in refractory or recurrent ascites.There are no reports on the use of combination of midodrine and tolvaptan in the patients with cirrhosis with ascites. Therefore, we plan to study the role of midodrine, tolvaptan and their combination on systemic hemodynamics, renal functions and control of ascites in patients with cirrhosis and refractory or recurrent ascites.

ELIGIBILITY:
Inclusion Criteria:60 consecutive patients with cirrhosis and refractory or recurrent ascites with stable renal function ( creatinine level <1.5mg/dl for at least 7 days ).

Exclusion Criteria:

* Presence of gastrointestinal bleeding, HRS, hepatic encephalopathy of grade 2 or higher or infection within 1 month preceding the study or during the study, presence of diabetes, intrinsic renal or cardiovascular disease or arterial hypertension on history and physical examination, abnormal urine analysis, chest radiograph or electrocardiogram, presence of hepatocellular carcinoma or portal vein thrombosis or treatment with drugs with known effects on systemic and renal hemodynamics within 7 days of inclusion .

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2013-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Number of patients with control of ascites | 3 months
  Control of ascites will be defined as:
  Complete: defined as the elimination of ascites Partial: presence of ascites not requiring paracentesis Failure: defined as persistence of ascites requiring paracentesis

SECONDARY OUTCOMES:
Number of patients with worsening of encephalopathy | 3 months
Number of patients with impairment of liver function | 3 months
Number of patients with variceal bleed | 3 months
Number of patients developing hepatorenal syndrome | 3 months
Number of patients with hypernatremia | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Virendra Singh, Study Chair — PGIMER, Chandigarh
Locations (1):
- Dept. of Hepatology, PGIMER, Chandigarh, Chandigarh, India

REFERENCES:
- [Derived] Rai N, Singh B, Singh A, Vijayvergiya R, Sharma N, Bhalla A, Singh V. Midodrine and tolvaptan in patients with cirrhosis and refractory or recurrent ascites: a randomised pilot study. Liver Int. 2017 Mar;37(3):406-414. doi: 10.1111/liv.13250. Epub 2016 Oct 2. PMID 27614145